CLINICAL TRIAL: NCT03895671
Title: OPEN LABEL PHASE 2 STUDY ON THE EFFICACY AND TOLERANCE OF A COMBINATION OF PONATINIB AND 5-AZACITIDINE IN CHRONIC MYELOGENOUS LEUKAEMIA IN ACCELERATED PHASE OR IN MYELOID BLAST CRISIS - PONAZA TRIAL
Brief Title: PONAZA : A COMBINATION OF PONATINIB AND 5-AZACITIDINE IN CHRONIC MYELOGENOUS LEUKAEMIA IN ACCELERATED PHASE OR IN MYELOID BLAST CRISIS
Acronym: PONAZA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Clinical coordinator, Versailles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P16/23 PONAZA
Record Dates: First submitted 2019-03-25; First posted 2019-03-29 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: CHRONIC MYELOGENOUS LEUKAEMIA IN ACCELERATED PHASE; CHRONIC MYELOGENOUS LEUKAEMIA IN MYELOID BLAST CRISIS
MeSH Terms: interventions — ponatinib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AP-CML (Experimental): Patient with Philadelphia chromosome positive CML in accelerated phase is defined by the presence of 15-29% blasts in peripheral blood (PB) or bone marrow (BM), ≥ 20% basophils in PB or BM, ≥ 30% blasts plus promyelocytes (with blasts <30%) in PB or BM, <100 x109/L platelets unrelated to therapy, or by clonal cytogenetics evolution (i.e., the presence of cytogenetic abnormalities other than the Philadelphia chromosome);
  Interventions: Drug: Ponatinib; Drug: Azacitidine
- MBC-CML (Experimental): Patient with Philadelphia chromosome positive CML in myeloid blast crisis is defined by the presence of ≥ 30% blasts in the bone marrow and/or peripheral blood or the presence of extramedullary disease.
  Interventions: Drug: Ponatinib; Drug: Azacitidine

INTERVENTIONS:
Drug: Ponatinib — Induction phase (first three cycles)
  - ponatinib: 45 mg/day orally continuously
  Following the results of disease evaluation after 3 cycles:
  * Cohort A: AP-CML If a CHR and complete cytogenetic response are obtained after 3 months, ponatinib will be decreased at 30mg/day. If CHR and/or CCyR are not reached, ponatinib may be maintained at 45mg/day for another 3 cycles if decided by the investigator.
  * Cohort B: MBC-CML If a CHR is obtained during the induction phase, ponatinib daily dose will be reduced to 30 mg/day. If CHR is not reached, ponatinib may be maintained at 45mg/day for another 3 cycles if decided by the investigator.
  Maintenance therapy:
  Ponatinib will be decreased to 30 mg/day. During maintenance therapy, If a major molecular response is reached, ponatinib will be decreased to 15mg/day
Drug: Azacitidine — Induction phase (first three cycles), Following the results of disease evaluation after 3 cycles and Maintenance therapy:
  - 5-azacitidine : 75 mg/m² subcutaneously day 1 to day 7, every 4 weeks
  No dose modification of 5-Azacitidine is planned in both cohorts. Azacitidine may be stopped at 24 months in case of MR4 defined as 0.0032%<MR4≤0.01%;

SUMMARY:
This project is strategy aiming to improve the survival of patients with chronic myelogenous leukemia in advanced phase and myeloid blast crisis.

The basis of this strategy is to add the demethylating agent 5-Azacitidine to the tyrosine kinase inhibitor ponatinib and evaluate its activity in 2 cohorts of patients with either chronic myelogenous leukemia in advanced phase or myeloid blast crisis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or more
2. Signed informed consent
3. Patient with Philadelphia chromosome positive CML in first blast crisis or first accelerated phase:

   * AP-CML is defined by the presence of any of the following features:

     * 15-29% blasts in peripheral blood (PB) or bone marrow (BM)
     * ≥ 20% basophils in PB
     * ≥ 30% blasts plus promyelocytes (with blasts <30%) in PB or BM,
     * <100 x10(9)/L platelets unrelated to therapy, or by clonal cytogenetics evolution (i.e., the presence of cytogenetic abnormalities other than the Philadelphia chromosome);
   * MBC-CML is defined by the presence of ≥ 30% blasts in the bone marrow and/or peripheral blood or the presence of extramedullary disease.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 or 3
5. Have adequate renal function as defined by the following criterion: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) for institution
6. Have adequate hepatic function as defined by the following criteria:

   1. Total serum bilirubin ≤ 1.5 × ULN, unless due to Gilbert's syndrome or CML
   2. Alanine aminotransferase (ALT) ≤ 2.5 × ULN, or ≤ 5 × ULN if leukemic infiltration of the liver is present
   3. Aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5 × ULN if leukemic infiltration of the liver is present
7. Have normal pancreatic status as defined by the following criterion: Serum lipase and amylase ≤ 1.5 × ULN
8. Have normal QTcF interval on screening electrocardiogram (ECG) evaluation, defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
9. Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
10. Agree to use an effective form of contraception with sexual partners throughout study participation (for female and male patients who are fertile).
11. Have fully recovered (≤ grade 1, returned to baseline, or deemed irreversible) from the acute effects of prior cancer therapy before initiation of study drug

Exclusion Criteria:

1. Pregnant or lactating women,
2. Participation in another clinical trial with any investigative drug within 30 days prior to study enrolment,
3. Prior history of hematopoietic stem cell transplantation
4. Cardiovascular disease:

   * Stage II to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system for heart failure.
   * Myocardial infarction within the previous 6 months
   * Symptomatic cardiac arrhythmia requiring treatment
5. Individuals with another active malignancy
6. Patients at high risk or very high risk of arterio-veinous occlusive disease defined by European CVD score
7. Previous treatment with azacitidine,
8. Diagnosis of malignant disease within the previous 12 months (excluding base cell carcinoma, "in-situ" carcinoma of the cervix or breast or other local malignancy excised or irradiated with a high probability of cure)
9. Known active viral infection with Human Immunodeficiency Virus (HIV) or Hepatitis type B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  To determine the overall survival of patients with AP-CML (cohort A) and MBC-CML (cohort-B) treated with the combination ponatinib and 5-azacitidine

SECONDARY OUTCOMES:
safety of combination of ponatinib and 5-azacitidine | 1 year
  To determine the safety of combination ofponatinib and 5-azacitidine: number adverse events related to ponatinib assessed by CTCAE V4.0
rate of Complete Hematologic Response (CHR) | 1 year
  To assess the rate of CHR : number de patient in complete hematologic response
cytogenetic response | 1 year
  To assess the complete cytogenetic response by caryotype analysis
molecular response | 1 year
  To assess the major molecular responseby BCR-ABL IS quantification
rate of reversion to chronic phase CML | 1 year
  To assess the rate of reversion to chronic phase CML
duration of response | 1 year
  To estimate the duration of response
duration of event free survival | 1 year
  To estimate the duration of event-free survival
relationship between clinical efficacy and biological markers (mutations and methylation status | 1 year
  To investigate the relationship between clinical efficacy and biological markers: mutations and methylation status.
allogenic transplant | 1 year
  To estimate the rate of patients bridged to allogenic transplant
Survival after transplant | 1 year
  To follow up event-free survival after transplant

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - Centre Hospitalier Universitaire D'Amiens, Amiens
  - Centre Hospitalier D'Avignon, Avignon
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Caen-Normandie, Caen
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hopital Pitie-Salpetriere, Paris
  - Hopital St Antoine, Paris
  - Hopital St Louis, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Hospices Civils de Lyon, Pierre-Bénite
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier de Strasbourg, Strasbourg
  - Institut Universitaire Du Cancer Toulouse, Toulouse
  - Chru de Nancy, Vandœuvre-lès-Nancy
  - Centre Hospitalier de Versailles, Versailles
  - Intitut Gustave Roussy, Villejuif